CLINICAL TRIAL: NCT02706964
Title: Imaging the Patterns of Breast Cancer Early Metastases
Acronym: BCMetPats
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Florida Academic Cancer Center Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201500683
Record Dates: First submitted 2016-03-07; First posted 2016-03-11 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: metastasis; 3D imaging; early detection
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Positron Emission Tomography Computed Tomography; Magnetic Resonance Imaging; Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proactive imaging (Experimental): All enrolled subjects will under go a single whole-body Positron emission tomography/x-ray computed tomography (PET/CT) scan and a diagnostic-quality x-ray computed tomography (CT) scan with contrast acquired in the same imaging session; and a single brain magnetic resonance imaging (MRI) scan with contrast to be completed in separate imaging session but within 2 weeks of the PET/CT scan. Imaging will take place within 7 months after enrollment.
  Interventions: Device: Positron emission tomography/x-ray computed tomography; Device: Magnetic resonance imaging; Device: x-ray computed tomography (CT)

INTERVENTIONS:
Device: Positron emission tomography/x-ray computed tomography — A whole-body PET/CT will be performed to identify the site and extent of spread.
  Other Names: PET/CT
Device: Magnetic resonance imaging — A brain MRI will be performed.
  Other Names: MRI
Device: x-ray computed tomography (CT) — A CT scan will be performed to identify the site and extent of spread.
  Other Names: CT

SUMMARY:
Currently, once a distant breast metastasis has been diagnosed, 65% of patients will succumb to their cancer within 2 years, and 80% will succumb by 5 years. The current National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Breast Cancer do not recommend surveillance imaging for earlier detection of distant metastases, even for high-risk breast cancer patients. Whereas, the standard-of-care treatment of the small isolated (few in number) breast cancer metastases is to perform surgical resection or locally ablative radiation therapy, however, the follow-up of breast cancer patients (including those with a >= 30% risk of developing metastases) is to wait for clinical symptoms to appear before using a dual positron emission tomography (PET) and diagnostic quality computed tomography (CT) PET/CT scan, magnetic resonance imaging (MRI), computed tomography (CT) or a bone scan to identify the site and extent of spread. Unfortunately, once metastases become symptomatic they are often too large and/or numerous to treat with curative intent. The current national care guidelines that advocate against intensive surveillance for distant metastases are based on two studies performed in Italy from 1985-1993 that concluded that the available imaging and treatment tools of the day did not prolong 5-year survival. Since then, however, there have been major improvements in imaging and treatment technology. To be treatable the metastases must be limited in number and limited in size, typically 6 or fewer metastases, each of size 5 centimeter or less. This state of metastatic presentation is called oligometastases. Numerous pilot studies have achieved dramatically improved overall and disease-free survival when oligometastases are treated using a combined systemic plus locally-ablative therapy of each oligometastasis. A scientific concern with the aforementioned research studies involving ablation of isolated oligometastases, was that they were not carried out with consistent use of surveillance imaging. Instead, these studies effectively preselected patients for enrollment based upon having an existing oligometastatic presentation. The primary objectives of the research study are to: (1) determine the feasibility of the stated interventions in a multi-institutional setting; (2) document the patterns of early metastatic spread of breast cancer; (3) document the proportion of high-risk breast cancer patients that have an oligometastatic presentation within this proactive imaging protocol, and (4) provide a basis to determine how to optimize future surveillance imaging protocols with respect to the time to progression, rate of tumor growth and organs that are affected.

DETAILED DESCRIPTION:
All enrolled subjects will undergo a single whole-body dual positron emission tomography (PET) and diagnostic quality computed tomography (CT) PET/CT scan and a CT scan with contrast acquired in the same imaging session; and a single brain magnetic resonance imaging (MRI) scan with contrast to be completed in separate imaging session but within 2 weeks of the PET/CT scan. Imaging will take place within 7 months after enrollment. In addition, the medical records related to the breast cancer and care, obtained and maintained as per standard-of-care, will be monitored for up to 5 years.

In this research study the investigators will acquire a PET/CT image of the body (neck to mid-thigh) using best-practice diagnostic imaging protocols, typically involving 64-slice CT systems, 1x1x3 mm voxel dimensions, use of non-ionic contrast agents, and breath-holding for motion correction. Subjects will also receive a single MRI with injected contrast of the brain using best-practice diagnostic imaging protocols, typically involving a 3-Tesla clinical MRI system.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with breast cancer who have completed radiation therapy within the last 48 months with a diagnosis that associates them with high risk (>30%) for developing metastatic disease but who at the time of enrollment are not known to have metastatic disease. Patients meeting this criterion are those that have either of the following presentations:
* hormone receptor (or triple) negative breast cancer with 3 or more positive axillary lymph nodes;
* a Stage III diagnosis;
* a primary tumor >2 cm and positive axillary lymph nodes;
* multiple primary tumors with cumulative volume >= that of a single 2 centimeter tumor, and positive axillary lymph nodes
* any number of lymph nodes with extranodal extension;
* any internal mammary or supraclavicular nodes;
* any primary tumor that has grown into the chest wall or skin;
* or inflammatory breast cancer.

Exclusion Criteria:

* Patients not willing to submit to a PET/CT scan and a brain MRI scan with injected vascular contrast at the Department of Radiology at University of Florida or University of Miami.
* Pregnant women are excluded because of possible radiation risk to the fetus.

Ages: 18 Years to 110 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with oligometastatic presentation | year 1
  Count the number of metastatic lesions at first imaging-incidence of presentation based on radiologist findings and application of the PI's computer-based automatic tumor detection program. If the number is 5 or less and none are > 5 cm in diameter, then this defines and oligometastatic presentation. Comparator: when metastases are first detected upon presentation of clinical symptoms, only 18% of patients are oligometastatic.
Histogram of the number and size of metastases at first presentation. | year 1
  Count of the number of metastases and their size based on radiologists findings and application of the PI's computer-based automatic tumor detection and sizing program. Goal to generate a histogram of tumor number and size.
Measure time to first instance of metastatic presentation. | year 1
  Record when the metastases are first discovered across the population of patient subjects.
Measure the growth rates of metastases in each of the target organs. | year 1
  Based on repeated follow-up scans we will use the PI's automated tumor sizing algorithm to computer tumor growth rates and compare growth rates across the different organs to which breast cancer spreads to (e.g., lung, liver, brain, spine).
Measure the incidence of metastatic spread to each target organ. | year 1
  Count of the number of metastases to each distant site, and their incidence, based on radiologists findings.
Prognosis for oligometastases based on patient and tumor factors. | year 1
  Measure primary breast tumor factors of size, number, type (ER/PR/HER2, luminal, basal), stage, nodal stage, etc., and patient factors of age, race, smoking history, etc. and correlate this in a multivariate analysis with the number of metastases at first presentation (including proportion of patients with oligometastases).

SECONDARY OUTCOMES:
Local control outcomes of treatment of metastases | Years 1-5
  In those patients who present with metastases under the imaging protocol and go on to receive additional treat of those metastases, to measure the local control rate and compare with historical controls.
Acute and late clinical side effects for ablative local therapy of the metastases | Years 1-5
  In those patients who present with metastases under the imaging protocol and go on to receive additional treat of those metastases, to measure clinical acute and late side-effects of treatment and compare with historical controls.
Patterns of secondary recurrence | Years 1-5
  Repeat each of the outcomes analyses above but for secondary instance of distant metastases instance, in those patients who receive treatment of breast cancer metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Walter G O'Dell, PhD, Principal Investigator — University of Florida, Assistant Professor of Radiation Oncology
Locations (2):
- United States (2):
  - Department of Radiation Oncology Davis Cancer Pavilion, Gainesville, Florida
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida

IPD SHARING:
Plan to Share IPD: No